CLINICAL TRIAL: NCT00020176
Title: Allogeneic Breast Protocol 1: T-Cell Depleted Allogeneic Blood Stem Cell Transplantation Using an Immunoablative Conditioning Regimen in Metastatic Breast Cancer
Brief Title: Allogeneic Peripheral Stem Cell Transplantation in Treating Patients With Stage IV Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000067899; NCI-00-C-0119; NCI-1027; NCT00005568 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2004-11

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer; male breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Filgrastim; Cyclophosphamide; Cyclosporine; fludarabine phosphate; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: filgrastim
Biological: therapeutic allogeneic lymphocytes
Drug: cyclophosphamide
Drug: cyclosporine
Drug: fludarabine phosphate
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Peripheral stem cell transplantation may be able to replace immune cells that were destroyed by chemotherapy used to kill tumor cells.

PURPOSE: Phase II trial to study the effectiveness of allogeneic peripheral stem cell transplantation in treating patients who have stage IV breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the ability of T-cell-depleted allogeneic blood stem cell transplantation after an immunoablative conditioning regimen to induce a state of mixed host/donor chimerism in patients with metastatic breast cancer.
* Determine the ability of this treatment regimen to induce an allogeneic graft-versus-tumor response in these patients.
* Determine the feasibility of giving other approved therapies to these patients at the first sign of disease progression in order to stabilize or produce a minimal or partial response.

OUTLINE: Patients receive chemotherapy comprising fludarabine IV over 30 minutes and cyclophosphamide IV over 1 hour on days 1-4. Patients receive filgrastim (G-CSF) SC daily beginning on day 5 and continuing until blood counts recover. Treatment repeats every 21 days for a maximum of 2 courses.

Patients receive a transplantation preparative regimen comprising fludarabine IV over 30 minutes and cyclophosphamide IV over 2 hours on days -6 to -3 (beginning on day 22 of immune-depleting chemotherapy) followed by allogeneic peripheral blood stem cell transplantation IV on day 0. Patients receive G-CSF SC daily beginning on day 0 and continuing until blood counts recover, plus cyclosporine IV over 1-2 hours every 12 hours on days -1 to 14 and then orally until day 40.

Patients with persistent malignant disease and less than grade II acute graft-versus-host disease receive donor lymphocytes IV on days 42, 70, and 98.

Patients are followed twice weekly until day 100, and then at 6, 9, 12, 18, and 24 months.

PROJECTED ACCRUAL: A maximum of 70 patients will be accrued for this study within 24 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Stage IV breast cancer
* Measurable disease
* Progressive disease

  * Increase in disease mass or less than partial response to therapy
  * At least one prior chemotherapy regimen for metastatic disease and progressed

    * Must have received prior therapy with a taxane and an anthracycline
* Estrogen/progesterone receptor-positive patients must have received and progressed on at least one hormonal agent in adjuvant or metastatic setting
* Her2-neu-expressing patients must have received and progressed on trastuzumab (Herceptin®) in adjuvant or metastatic setting
* Prior autologous stem cell transplantation allowed if less than complete response or disease progression in adjuvant or metastatic setting
* Consenting first-degree relative with at least 5 out of 6 HLA-antigen match (may include mismatch at the D locus)
* Hormone receptor status:

  * Estrogen receptor status known
  * Progesterone receptor status known

PATIENT CHARACTERISTICS:

Age:

* 18 to 70

Sex:

* Male or female

Menopausal status:

* Not specified

Performance status:

* Karnofsky 80-100%

Life expectancy:

* More than 6 months

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin ≤ 2 mg/dL
* SGOT < 4 times upper limit of normal
* Hepatitis B surface antigen negative
* Hepatitis C antibody negative

Renal:

* Creatinine ≤ 1.5 mg/dL
* Creatinine clearance ≥ 50 mL/min

Cardiovascular:

* Left ventricular ejection fraction > 45%

Pulmonary:

* DLCO ≥ 50% of predicted

Other:

* HIV negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics
* Recovered from prior stem cell transplantation

Chemotherapy:

* See Disease Characteristics

Endocrine therapy:

* See Disease Characteristics
* No concurrent steroids

Radiotherapy:

* Not specified

Surgery:

* Not specified

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-06; Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael R. Bishop, MD, Principal Investigator — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - NCI - Center for Cancer Research, Bethesda, Maryland

REFERENCES:
- [Background] Bishop MR. Nonmyeloablative allogeneic hematopoietic stem cell transplantation for metastatic breast cancer. Clin Breast Cancer. 2003 Apr;4(1):39-45. doi: 10.3816/cbc.2003.n.010. PMID 12744757
- [Result] Bishop MR, Fowler DH, Marchigiani D, Castro K, Kasten-Sportes C, Steinberg SM, Gea-Banacloche JC, Dean R, Chow CK, Carter C, Read EJ, Leitman S, Gress R. Allogeneic lymphocytes induce tumor regression of advanced metastatic breast cancer. J Clin Oncol. 2004 Oct 1;22(19):3886-92. doi: 10.1200/JCO.2004.01.127. Epub 2004 Aug 16. PMID 15314059
- [Result] Bishop MR, Steinberg SM, Gress RE, Hardy NM, Marchigiani D, Kasten-Sportes C, Dean R, Pavletic SZ, Gea-Banacloche J, Castro K, Hakim F, Krumlauf M, Read EJ, Carter C, Leitman SF, Fowler DH. Targeted pretransplant host lymphocyte depletion prior to T-cell depleted reduced-intensity allogeneic stem cell transplantation. Br J Haematol. 2004 Sep;126(6):837-43. doi: 10.1111/j.1365-2141.2004.05133.x. PMID 15352988
- [Result] Bishop MR, Kasten-Sportes C, Dean R, et al.: Preemptive DLI after T cell-depleted reduced-intensity allogeneic HSCT for metastatic breast cancer: effect on engraftment, GVHD, and anti-tumor response. [Abstract] Blood 102 (11): A- 5567, 2003.
- [Result] Bishop MR, Marchigiani D, Grasmeder S, et al.: Demonstration of clinical responses to adoptive cellular therapy using allogeneic T cells in metastatic breast cancer. [Abstract] Proceedings of the American Society of Clinical Oncology 22: A-657, 2003.
- [Result] Bishop MR, Marchigiani D, Odom J, et al.: Contribution of T cells to engraftment: a comparison of T cell depleted vs. T cell replete allografts after reduced-intensity conditioning. [Abstract] Blood 102 (11): A-2447, 2003.